CLINICAL TRIAL: NCT03190226
Title: L-PRF Membranes for Increasing the Width of Keratinised Mucosa Around Implants: A Split-mouth, Randomized, Controlled Pilot Clinical Trial
Brief Title: L-PRF for Increasing Keratinised Mucosa Around Implants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S57225
Record Dates: First submitted 2017-05-29; First posted 2017-06-16 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2016-05

CONDITIONS: Implantation Complication
Keywords: L-PRF; keratinised tissues; implant; free gingival graft

STUDY DESIGN:
Intervention Model Description: split-mouth trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- L-PRF membranes (Experimental): Intra-oral split thickness preparation - apically repositioned to the periosteum.
  L-PRF membranes will be used to cover the site. Free Gingival Grafts will be used to cover the site.
  Interventions: Procedure: L-PRF membranes; Procedure: Free Gingival Graft

INTERVENTIONS:
Procedure: L-PRF membranes — split-mouth design, randomized L-PRF membranes vs. free gingival graft
Procedure: Free Gingival Graft — split-mouth design, randomized L-PRF membranes vs. free gingival graft

SUMMARY:
The aim of this study was to evaluate the potential of L-PRF in increasing the width of the keratinsed mucosa around implants. Furthermore, it was assessed whether this surgery was associated with significantly less post-operative discomfort for the patient compared to Free Gingival Graft surgery. L-PRF for increasing keratinised mucosa around implants.

ELIGIBILITY:
Inclusion Criteria:

* in need of bilateral enlargement of keratinsed tissues around implants

Exclusion Criteria:

* smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-27 (Actual); Study Completion 2017-05-27 (Actual)

PRIMARY OUTCOMES:
Amount of keratinised tissues | Measurements were performed pre-operatively (using lugol staining) and 3 months after surgery (using lugol staining). Results will be presented in the final paper.
  measurements of changes in amount of keratinised tissues

SECONDARY OUTCOMES:
Post-op pain assessment | Visual analogue scales were handed out after surgery and were collected 1 week post-operatively. Results will be presented in the final paper.
  Post-operative pain assessment via VAS-scales

CONTACTS AND LOCATIONS:
Overall Officials: Gert-Jan Cleeren, MSc, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No